CLINICAL TRIAL: NCT05462249
Title: Impact of Catch-up HPV Vaccination on the Development of Cervical Lesions
Brief Title: Impact of Catch-up HPV Vaccination
Acronym: HPVAC2
Status: Terminated | Type: Observational
Why Stopped: overestimation of the number of healthcare professionals participating in the inclusions
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: HPVAC2 - 29BRC21.0008
Record Dates: First submitted 2022-07-07; First posted 2022-07-18 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: HPV; HPV Vaccination; Vaccine Preventable Disease; Cervical Lesion; Cervical Cancer
MeSH Terms: conditions — Vaccine-Preventable Diseases; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Vaccinated: Patients who have been vaccinated against HPV virus.
- Not vaccinated: Patients who have not been vaccinated against HPV virus.

SUMMARY:
Each year in France, more than 6000 new cases of HPV inducted cancers are recorded. The vaccinal cover stays insufficient since less than 30% of the french population is vaccinated. Therefore french studies about vaccine efficacy and especially about the catch-up vaccine (done after 15years old) are needed.

HPVAC2 is a prospective, analytic and monocentric study designed to learn the impact of the catch-up HPV vaccination.

Women from 25 years old and born after 1984 may be included if they come to the Brest CHU to do their regular cervical smear. At this time, a survey will be given to know their vaccinal status.

The aim of the study is to prove the efficacy of the catch up vaccination by analyzing the cervical smears results and by comparing the vaccinated group with the not-vaccinated group.

ELIGIBILITY:
Inclusion Criteria:

* Age limit
* Patient must have done a HPV or smear test during the study period
* Consent necessary

Exclusion Criteria:

* Age limit
* No HPV or smear test done in the study period
* Patient not able to give her consent

Ages: 25 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women between 25 and 38 years old in 2022 coming for a HPV or smear test during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 354 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Test HPV and smear test result. | 13 months.
  Study the effectiveness of anti-HPV vaccine (done between 15 and 19 years old).

SECONDARY OUTCOMES:
Test HPV and smear test result. | 13 months.
  Study the effectiveness of anti-HPV vaccine (done between 11 and 15 years old).
Test HPV and smear test result. | 13 months.
  Study the effectiveness of anti-HPV vaccine (not regarding the period of realization)
Test HPV and smear test result. | 13 months.
  Compare the effectiveness of anti-HPV vaccine done before and after 15 years old.
Test HPV and smear test result regarding the cervical cancer risk factors. | 13 months.
  Study the impact of the known cervical cancer risk factors on the smear results.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe MERVIEL, PU-PH, Study Director — Head of the gynecologic department in Brest Hospital
Locations (1):
- CHU de BREST, Brest, Finistère, France

IPD SHARING:
Plan to Share IPD: No
All the data are anonymized.